CLINICAL TRIAL: NCT06326372
Title: The Effect of Intraoperative Hyperoxemia on Postoperative Delirium in Geriatric Patients and the Preventive Role of Oxygen Reserve Index"
Brief Title: The Effect of Intraoperative Hyperoxemia on Postoperative Delirium in Geriatric Patients
Status: Completed | Type: Observational
Sponsor: Tepecik Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Aykut Saritas, associated professor, Tepecik Training and Research Hospital
Other Study IDs: Delirium
Record Dates: First submitted 2024-03-16; First posted 2024-03-22 (Actual); Last update posted 2024-07-09 (Actual); Status verified 2024-03

CONDITIONS: Hyperoxia; Delirium in Old Age
MeSH Terms: conditions — Hyperoxia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Control group: In the control group, observation will be conducted solely by another anesthesia doctor or assistant participating in the study, and the data will be recorded blindly without being reported to the anesthesia doctor responsible for the surgery. The oxygen therapy administered by the anesthesia doctor in charge and the FiO2 values will be recorded independently and blindly, based solely on the clinician's own assessment, rather than according to the information obtained from ORi. Subsequently, for two days following the surgery, evaluations will be conducted twice daily at the same hours for ward patients using CAM, and for ICU patients using CAM-ICU. If delirium is detected, delirium subtyping will be performed using the Richmond Agitation-Sedation Scale (RASS).
  Interventions: Procedure: control
- ORi+SpO2 group: In the SpO2+ORi group; It is aimed to maintain SpO2 between %95 and %98, and ORi at 0.00.
  Data will be recorded every 10 minutes. After extubation, patients will first be evaluated in the postoperative recovery room. Subsequently, for two days following the surgery, evaluations will be conducted twice daily at the same hours for ward patients using CAM, and for ICU patients using CAM-ICU. If delirium is detected, delirium subtyping will be performed using the Richmond Agitation-Sedation Scale (RASS).
  Interventions: Procedure: ORi+SpO2

INTERVENTIONS:
Procedure: control — Fraction of inspired oxygen (FiO2) is titrated guided by oxygen saturation in that range; %95<oxygen saturation
  Groups: Control group
Procedure: ORi+SpO2 — Titration of fraction of inspired oxygen (FiO2) guided by ORI and oxygen saturation FiO2 will be titrated by reducing 10% if Ori>0.01 and oxygen saturation ≥ 98% until Ori is 0.00.
  FiO2 will not be changed if Ori is 0.00 and %95<oxygen saturation≤%98 FiO2 will be increased by 10% if oxygen saturation <95 or PaO2<60 mmHg
  Groups: ORi+SpO2 group

SUMMARY:
Oxygen therapy is the most common treatment modality for patients with hypoxemia, but target values for normoxemia are not clearly defined. Therefore, iatrogenic hyperoxemia is a very common situation. Even though there are many side effects reported related to hyperoxemia and hyperoxemia is shown to be related to worse outcome than expected; clinicians still observe hyperoxemia frequently.

Oxygen reserve index (ORi™) (Masimo Corp., Irvine, USA) can guide clinicians in detection of hyperoxia. ORi is a parameter which can evaluate partial pressure of oxygen (PaO2) rating from 0 to 1. There are growing evidences in ORi that it might be helpful to reduce hyperoxia in general anesthesia. Continuous ORi monitoring can be used for detecting and preventing hyperoxia. The ability to perform FiO2 titration with ORi may be an appropriate monitoring management to prevent the harmful effects of hyperoxia.In this study, in patients who underwent major abdominal surgery; It was aimed to investigate the effectiveness of ORi-guided FiO2 titration in preventing hyperoxia.

DETAILED DESCRIPTION:
The definition of elderly by the World Health Organization is individuals aged 65 and older. As the average life expectancy continues to increase, the number of surgical procedures performed in the geriatric population is also increasing.

Postoperative delirium is a complication that occurs after surgery and is characterized by sudden-onset confusion, fluctuating mental status, and attention deficits. Its incidence increases in elderly patients and is higher in those with pre-existing mild cognitive impairment. The etiology encompasses multiple factors such as age, presence of additional comorbidities, metabolic disorders, hypoxia, polypharmacy, pain, hypothermia, and may be associated with the depth of anesthesia during surgery.

Early recognition and prevention of delirium will become more prominent in the future due to reduced hospitalization durations, postoperative complications, and mortality rates.

Various methods are available to detect hyperoxemia during surgery. Hyperoxemia can be detected using noninvasive finger pulse oximetry with the oxygen reserve index parameter. Oxygen levels can be noninvasively assessed during operations using routine oxygen saturation and oxygen reserve index measurements.

Delirium can be evaluated in both intensive care and ward patients. The gold standard for diagnosis is the Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-5) criteria. DSM-5 criteria require psychiatric evaluation and are conducted by someone with psychiatric training. Additionally, the Confusion Assessment Method (CAM) is used for diagnosis and can be evaluated as CAM-ICU for intubated patients in intensive care units.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged 65 and older
2. Patients expected to have surgery lasting more than 2 hours
3. Patients with ASA (American Society of Anesthesiologists) classification 1-2-3-4
4. Patients planned to have at least 2 days of postoperative hospitalization

Exclusion Criteria:

1. Patients with preoperative central nervous system disorders or dementia
2. Patients with MMSE (Mini-Mental State Examination) scores of 23 or below
3. Patients unable to communicate
4. Emergency surgeries
5. Patients who refuse to participate in the study
6. Patients using high-dose vasopressors
7. Patients with peripheral hypoperfusion
8. Hemodynamically unstable patients

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: Patients aged 65 and older. Geriatric patients
Sampling Method: Probability Sample
Enrollment: 114 (Actual)
Dates: Start 2023-10-01 (Actual); Primary Completion 2024-07-05 (Actual); Study Completion 2024-07-07 (Actual)

PRIMARY OUTCOMES:
Correlation of FiO2 and ORi value | Until the surgery is over
  Correlation of FiO2 value and ORi value. FiO2 adjusted until ORi reaches to zero and %95<oxygen saturation≤%98
Correlation of ORi and Delirium | Up to 48 hours
  Correlation of ORİ and SpO2 values with delirium measured by CAM and CAM-ICU

SECONDARY OUTCOMES:
Correlation of FiO2 and delirium | first 10 th minutes after entubation and every 10 minutes until surgery is over
  Correlation of FiO2 and delirium measured by CAM and CAM-ICU

CONTACTS AND LOCATIONS:
Locations (1):
- Aykut Saritaş, Izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided